CLINICAL TRIAL: NCT01370759
Title: Flocculation-Adsorption System for Colon Cleansing Enhancement: A Feasibility Study
Brief Title: Feasibility Study to Evaluate the Performance of Flocculation-Adsorption System for Colon Cleansing Enhancement
Acronym: RD-400
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to sponsor desicioun
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CTIL - RD-400
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2014-04

CONDITIONS: Healthy
Keywords: bowel prep; PillCam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colon-targeted cleaning capsule (Experimental)
  Interventions: Other: Cleaning capsule

INTERVENTIONS:
Other: Cleaning capsule — Capsules containing the tested materials aimed to improve colon cleansing
  Other Names: Active cleaning capsules

SUMMARY:
The purpose of this study is to demonstrate feasibility of enhancing colon cleansing.

DETAILED DESCRIPTION:
To ensure the success of a PillCamTM Colon examination, as standard practice, patients are requested to adhere to a bowel preparation procedure.

The study is designed to evaluate the performance and contribution of a flocculation-adsorption system to colon cleansing.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age is between 23-75 years.
* Subject is healthy.
* Subject agrees to sign the Informed Consent Form

Exclusion Criteria:

* Contraindication to capsule endoscopy
* Contraindication or allergy to any of the products and materials used for bowel preparation
* Subject is not able to provide written informed consent

Ages: 23 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cleansing grading | within 10 days

SECONDARY OUTCOMES:
Distribution of time | within 10 days
GI tract segment of capsule disintegration | within 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gralnek, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical center, Haifa, Israel